CLINICAL TRIAL: NCT00232921
Title: The Effect of Caudal Volumes on the Anatomical Spread of Caudals in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 02AR07
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Asa 1 and 2 Patients for Elective Surgery Requiring Caudal as Part of Their Care

INTERVENTIONS:
Drug: caudal volume 1
Biological: caudal volume 2
Drug: caudal volume 3

SUMMARY:
Radiological study into the anatomical spread of caudal local anaesthetic in children age 1-7

ELIGIBILITY:
Inclusion Criteria:

* Asa 1 and 2 patients

Exclusion Criteria:

-

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 2003-02

PRIMARY OUTCOMES:
The radiographic height of the block post injection

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thomas, Dr, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom